CLINICAL TRIAL: NCT00139477
Title: Understanding the Effects of Therapeutic Intervention on Cardiovascular Risk Markers, Insulin Resistance, and Intra-Hepatic Fat Contents in Obese Children at High Risk for the Metabolic Syndrome.
Brief Title: Study of Serum Markers for Cardiovascular Risk in Obese Youth and Impact of Lifestyle and Medication Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Nelly Mauras, Principal investigator, Nemours Children's Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 04-032
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2012-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Metformin; Diet Therapy; Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diet/Exercise only, then Diet/Exercise plus Metformin (Experimental): Diet/Exercise only in first intervention period and Diet/Exercise plus Metformin in second intervention period (no washout period).
  Interventions: Drug: Metformin; Behavioral: Dietary modification with caloric restriction; Behavioral: Establishment of exercise protocol
- Diet/Exercise plus Metformin, then Diet/Exercise only (Active Comparator): Diet/Exercise plus Metformin in first intervention period and Diet/Exercise only in second intervention period (no washout period).
  Interventions: Drug: Metformin; Behavioral: Dietary modification with caloric restriction; Behavioral: Establishment of exercise protocol

INTERVENTIONS:
Drug: Metformin — Metformin, 250mg by mouth twice a day with meals will be started and if tolerated increased to 500mg twice a day in 3 days in those less than 12 years old and titrated further to 1000mg twice a day if tolerated.
Behavioral: Dietary modification with caloric restriction — The life style intervention changes will include a hypocaloric diet representing at least a 500 kcal/day reduction based on their dietary histories and Resting Energy Expenditure (REE) determined by the initial calorimetry.
Behavioral: Establishment of exercise protocol — Participants will attend the Fitness Center 3 times per week and supervised by an exercise technician or exercise specialist. Exercise will be individually prescribed for each participant based on their functional abilities. Exercise will consist of 5-10 minutes for warm up and stretching, followed by 15-30 minutes of cardiovascular exercise (i.e. treadmill, bicycle ergometer, rower, nustep, etc), 10-20 minutes of strength training (supervised using weight stack equipment), and 5-10 minutes of cool down and stretching. As children typically do not need an exercise prescription based on heart rate, we will familiarize them with perceived exertion scales and monitor that they are exercising in the moderate to hard range of perception of effort. Participants will be started at 15 minutes of cardiovascular exercise and 10 minutes of strength training exercise, progressing by 2-3 minutes every week until 30 and 20 minutes is achieved for each respectively.

SUMMARY:
In Protocol #2, we will select 30 obese pubertal and 30 obese prepubertal subjects with an abnormal cytokine profile (i.e. fibrinogen and/or hsCRP concentration greater than or equal to 2 Standard Deviations (SD) above the mean established in our lab for lean controls in Protocol #1). They will be randomly assigned to either lifestyle intervention (diet/exercise) or diet/exercise plus metformin for 6 months. After the 6 month evaluation the subjects will cross over the treatment arms, i.e., those that were doing diet/exercise intervention only will add metformin, those that were doing the diet/exercise plus metformin will discontinue the metformin and continue with diet/exercise changes only. Intrahepatic fat contents will be measured as well.

The investigators hypothesize that obese children in these age groups will have increased cardiovascular risk related to their obese state before reaching the currently defined criteria of metabolic syndrome.

The investigators hypothesize that these cardiovascular risks can be reduced with lifestyle and drug interventions.

ELIGIBILITY:
Inclusion Criteria:

* Ages 7-18 years.
* Greater than the 95th percentile body mass index for their age and gender.
* Children are in Tanner Stage I or IV or V.
* Normal Blood Pressure.
* Normal fasting glucose.
* Normal lipids.
* Menstruating girls must have completed their most recent period at least 2 weeks prior to blood draw.
* No recent illness, no chronic illnesses, no routine medications, no smoking or alcohol intake.
* Must pass the screening test done in Protocol #1.
* Must have higher values than normal for certain blood tests related to heart disease that were measured in Protocol #1.

Exclusion Criteria:

* Chronic active illnesses.
* Recent illnesses.
* Use of routine medications, vitamins, herbal remedies, oral contraceptive pills, or other over the counter medications within 4 weeks of blood draw.
* History of recent or chronic smoking.
* Currently pregnant.
* Impaired fasting glucose.
* Dyslipidemia.
* Actively in puberty.
* Weight greater than 300 pounds.
* Metal in the abdomen.
* History of being overweight greater than 5 years.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2003-11; Primary Completion 2009-05 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Mauras, MD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Result] Mauras N, Delgiorno C, Kollman C, Bird K, Morgan M, Sweeten S, Balagopal P, Damaso L. Obesity without established comorbidities of the metabolic syndrome is associated with a proinflammatory and prothrombotic state, even before the onset of puberty in children. J Clin Endocrinol Metab. 2010 Mar;95(3):1060-8. doi: 10.1210/jc.2009-1887. Epub 2010 Jan 8. PMID 20061420
- [Result] Rynders C, Weltman A, Delgiorno C, Balagopal P, Damaso L, Killen K, Mauras N. Lifestyle intervention improves fitness independent of metformin in obese adolescents. Med Sci Sports Exerc. 2012 May;44(5):786-92. doi: 10.1249/MSS.0b013e31823cef5e. PMID 22015710
- [Result] Mauras N, DelGiorno C, Hossain J, Bird K, Killen K, Merinbaum D, Weltman A, Damaso L, Balagopal P. Metformin use in children with obesity and normal glucose tolerance--effects on cardiovascular markers and intrahepatic fat. J Pediatr Endocrinol Metab. 2012;25(1-2):33-40. doi: 10.1515/jpem-2011-0450. PMID 22570948
- [Derived] Benson M, Hossain J, Caulfield MP, Damaso L, Gidding S, Mauras N. Lipoprotein subfractions by ion mobility in lean and obese children. J Pediatr. 2012 Dec;161(6):997-1003. doi: 10.1016/j.jpeds.2012.05.060. Epub 2012 Jul 20. PMID 22819275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from pediatric endocrinology clinics, in Jacksonville, USA between November 2003 and April 2008.
Pre-assignment Details: 375 participants recruited; 177 obese participants screened, 111 excluded (62 did not meet inclusion criteria and 4 refused participation).
Period: First Intervention -Baseline to 6Months
Arm/Group | Diet/Exercise Only, Then Diet/Exercise Plus Metformin | Diet/Exercise Plus Metformin, Then Diet/Exercise Only
Started | 31 | 35
Completed | 19 | 23
Not Completed | 12 | 12
Not completed — No Longer Interested | 6 | 7
Not completed — Relocation | 1 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Impaired Glucose Tolerance at Screening | 2 | 0
Period: Second Intervention -6Months to 12Months
Arm/Group | Diet/Exercise Only, Then Diet/Exercise Plus Metformin | Diet/Exercise Plus Metformin, Then Diet/Exercise Only
Started | 19 | 23
Completed | 14 | 18
Not Completed | 5 | 5
Not completed — No Longer Interested | 0 | 2
Not completed — Relocation | 1 | 0
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diet/Exercise Only, Then Diet/Exercise Plus Metformin | Diet/Exercise Plus Metformin, Then Diet/Exercise Only | Total
Number analyzed (Participants) | 31 | 35 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 35 | 66
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12 (0.4) | 12.3 (0.5) | 12.2 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  United States | 31 | 35 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in High-sensitivity C-reactive Protein (hsCRP) at 6 Months
Description: Value at 6 months minus value at baseline. HsCRP is an acute phase protein which is a sensitive marker for systemic inflammation. HsCRP concentrations were measured in our laboratory by immuno-nephelometry (Siemens Healthcare Diagnostics, Deerfield IL, USA), with an hsCRP lower sensitivity of 0.156 mg/L.
Time Frame: Baseline and 6 months
Population: 1 Subject in the "Diet/Exercise plus Metformin, then Diet/Exercise (Pubertal)" Group did not have an hsCRP level available for analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Groups:
- Diet/Exercise, Then Diet/Exercise Plus Metformin (Prepubertal); Diet/Exercise, Then Diet/Exercise Plus Metformin (Pubertal): Diet/Exercise only in first intervention period and Diet/Exercise plus Metformin in second intervention period (no washout period). Results displayed for prepubertal versus pubertal participants.
- Diet/Exercise Plus Metformin, Then Diet/Exercise (Prepubertal); Diet/Exercise Plus Metformin, Then Diet/Exercise (Pubertal): Diet/Exercise plus Metformin in first intervention period and Diet/Exercise only in second intervention period (no washout period). Results displayed for prepubertal versus pubertal participants.
Arm/Group | Diet/Exercise, Then Diet/Exercise Plus Metformin (Prepubertal) | Diet/Exercise, Then Diet/Exercise Plus Metformin (Pubertal) | Diet/Exercise Plus Metformin, Then Diet/Exercise (Prepubertal) | Diet/Exercise Plus Metformin, Then Diet/Exercise (Pubertal)
Number analyzed (Participants) | 8 | 11 | 13 | 9
mg/dL | -0.37 [-1.54 to 0.81] | -1.78 [-5.49 to -0.15] | -0.29 [-1.42 to 1.79] | 0.00 [-0.65 to 2.17]

2. Primary Outcome: Change From Baseline in Fibrinogen at 6 Months
Description: Value at 6 months minus value at baseline. Fibrinogen is a hepatic-derived factor directly involved in clotting and in the viscosity characteristics of blood flow. It binds to platelets and contributes to their aggregation, promotes fibrin formation and is also an acute phase reactant that is increased in inflammatory states. Fibrinogen concentrations were measured in our laboratory by immuno-nephelometry (Siemens Healthcare Diagnostics, Deerfield IL, USA).
Time Frame: Baseline and 6 months
Population: 1 Subject in the "Diet/Exercise plus Metformin, then Diet/Exercise (Pubertal)" Group did not have a Fibrinogen level available for analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Diet/Exercise, Then Diet/Exercise Plus Metformin (Prepubertal) | Diet/Exercise, Then Diet/Exercise Plus Metformin (Pubertal) | Diet/Exercise Plus Metformin, Then Diet/Exercise (Prepubertal) | Diet/Exercise Plus Metformin, Then Diet/Exercise (Pubertal)
Number analyzed (Participants) | 8 | 11 | 13 | 9
mg/dL | 58.5 [-64 to 123.75] | -105 [-141 to -31] | 0.00 [-51.5 to 83] | -33 [-93.5 to 40.5]

3. Primary Outcome: Change From Baseline in Interleukin 6 (IL-6) at 6 Months
Description: Value at 6 months minus value at baseline. IL-6 is a pro-inflammatory cytokine thought to produce a state of low-grade inflammation in obese individuals. IL-6 stimulates hepatic production of C-reactive protein (CRP), an acute phase protein which is a sensitive marker for systemic inflammation. IL-6 was measured by enzyme-linked immunosorbent assay (ELISA; R&D Systems, Minneapolis, MN, USA).
Time Frame: Baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Diet/Exercise, Then Diet/Exercise Plus Metformin (Prepubertal) | Diet/Exercise, Then Diet/Exercise Plus Metformin (Pubertal) | Diet/Exercise Plus Metformin, Then Diet/Exercise (Prepubertal) | Diet/Exercise Plus Metformin, Then Diet/Exercise (Pubertal)
Number analyzed (Participants) | 8 | 11 | 13 | 10
pg/mL | -0.66 [-2.39 to -0.01] | -0.99 [-2.11 to 0.22] | 0.2 [-0.80 to 2.19] | -0.35 [-0.94 to 0.07]

4. Primary Outcome: Change From Baseline in Plasminogen Activator Inhibitor-1 (PAI-1) at 6 Months
Description: Value at 6 months minus value at baseline. PAI-1 is the primary physiological inhibitor of fibrinolysis and proteolysis. High PAI-1 levels have been linked to thrombosis and fibrosis, insulin resistance and obesity. PAI-1 was measured by ELISA (American Diagnostica, Stamford, CT, USA).
Time Frame: Baseline and 6 months
Population: 1 Subject in the "Diet/Exercise plus Metformin, then Diet/Exercise (Pubertal)" Group and 1 Subject in the "Diet/Exercise, then Diet/Exercise plus Metformin (Pubertal)" Group did not have a PAI-1 level available for analysis.
Measure: Median (Inter-Quartile Range); unit: ng/ML
Arm/Group | Diet/Exercise, Then Diet/Exercise Plus Metformin (Prepubertal) | Diet/Exercise, Then Diet/Exercise Plus Metformin (Pubertal) | Diet/Exercise Plus Metformin, Then Diet/Exercise (Prepubertal) | Diet/Exercise Plus Metformin, Then Diet/Exercise (Pubertal)
Number analyzed (Participants) | 8 | 10 | 13 | 9
ng/ML | 6.98 [-48.54 to 14.4] | -46.84 [-62.86 to -24.46] | 0.55 [-34.45 to 34.22] | -34.42 [-46.74 to 25.82]

ADVERSE EVENTS:
Arm/Group | Diet/Exercise Only, Then Diet/Exercise Plus Metformin | Diet/Exercise Plus Metformin, Then Diet/Exercise Only
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/35
Other Adverse Events (participants affected / at risk) | 0/31 | 0/35

LIMITATIONS AND CAVEATS:
Protocol #2 attrition was high, such that, we could not derive conclusions beyond the 6 month time period. Therefore, conclusions were based on participants after completing the first intervention without crossover to the second intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes